CLINICAL TRIAL: NCT05946538
Title: Clinical Evaluation of SARS-COV-2, Influenza and RSV 8-Well MT-PCR Panel for In Vitro Diagnostics
Brief Title: Clinical Evaluation of SARS-COV-2 (COVID-19), Influenza and RSV 8-Well MT-PCR Panel for In Vitro Diagnostics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AusDiagnostics Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AUS-RES-01
Record Dates: First submitted 2023-07-12; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Respiratory Viral Infection
Keywords: In vitro Diagnostic Device; In vitro Diagnostic; Multiplexed Tandem Polymerase Chain Reaction; Respiratory Panel; Respiratory Syncytial Virus; Severe Acute Respiratory Syndrome Coronavirus 2; Influenza Virus

STUDY DESIGN:
Intervention Model Description: Prospective accuracy observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Device accuracy observational arm (Other): Two nasopharyngeal swabs will be collected from each enrolled participant and analysed on the AusDiagnostics in vitro diagnostic device panel and the comparator BioFire in vitro diagnostic device panel.
  Interventions: Diagnostic Test: SARS-COV-2, Influenza and RSV 8-Well MT-PCR Panel; Diagnostic Test: BioFire Respiratory Panel 2.1

INTERVENTIONS:
Diagnostic Test: SARS-COV-2, Influenza and RSV 8-Well MT-PCR Panel — The SARS-CoV-2, Influenza and RSV PCR test is multiplex-tandem polymerase chain reaction (MT-PCR) based on qualitive in vitro diagnostic testing for the detection and identification of pathogens in nucleic acid extracts.
Diagnostic Test: BioFire Respiratory Panel 2.1 — The BioFire Respiratory Panel 2.1 (RP2.1) is a PCR-based multiplexed nucleic acid test intended for use with the BioFire® FilmArray® 2.0 or BioFire® FilmArray® Torch Systems for the simultaneous qualitative detection and identification of multiple respiratory viral and bacterial nucleic acids in nasopharyngeal swabs (NPS) obtained from individuals suspected of respiratory tract infections.

SUMMARY:
This study is a prospective accuracy observational study to evaluate the performance of the Highplex System SARS-Cov-2, Influenza and RSV 8-well in vitro diagnostic medical device panel and generate performance data. The precision of results will be evaluated in concordance with the comparator predicate device panel BioFire Respiratory Panel 2.1 (RP2.1).

DETAILED DESCRIPTION:
This study is a prospective accuracy observational study to evaluate the performance of the Highplex System SARS-Cov-2, Influenza and RSV 8-well in vitro diagnostic medical device panel and generate performance data. The precision of results will be evaluated in concordance with the comparator predicate device panel BioFire Respiratory Panel 2.1 (RP2.1). This study will utilise prospective sample respiratory swabs from individuals with paired test data, presenting with influenza-like symptoms (e.g., cough, nasal congestion, rhinorrhoea, sore throat, fever, headache, myalgia), as well as asymptomatic individuals. To meet the target number of 400 positive samples (50 samples per target; 8 targets in total), a required sampling size of 1000 participants will need to be screened to account for unviable samples and screen failures. Prospective respiratory samples will include nasopharyngeal swabs as described in Intended Use of the product.

ELIGIBILITY:
Inclusion Criteria:

* The sample is derived from an individual who has the ability to provide consent or from a legally acceptable representative, parent(s), or legal guardian and have consented for their sample and demographic information to be taken
* The sample is a nasopharyngeal swab
* The sample is collected in universal transport media (UTM) or viral transport media (VTM), using FDA approved swabs
* The sample is collected from an individual who has a presumptive diagnosis or is presenting with influenza-like symptoms (e.g., cough, nasal congestion, rhinorrhoea, sore throat, fever, headache, myalgia) or is suspected to be asymptomatic.

Exclusion Criteria:

* Sample does not meet acceptable specimen criteria in that is not a nasopharyngeal swab
* The sample is collected using swabs with wood shafts or other materials known to inhibit growth of influenza viruses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with positive samples as evaluated by the AusDiagnostics SARS-COV-2, Influenza and RSV 8-Well MT-PCR Panel and the BioFire Respiratory Panel 2.1. | 6 months
  The study will be considered to have reached its primary endpoint when performance data from 50 positive samples for each panel target has been collected and evaluated for precision and concordance with the comparator predicate device panel BioFire Respiratory Panel 2.1 (RP2.1).